CLINICAL TRIAL: NCT02620540
Title: Evaluation of an Algorithm for Length Based Weight Estimation in Comparison to Already Known Devices Like the Broselow Tape (BT)
Brief Title: Evaluation of an Algorithm for Length Based Weight Estimation in Comparison to Known Devices
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0191 - Part 2
Record Dates: First submitted 2015-11-17; First posted 2015-12-03 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Weight-Estimation
Keywords: Broselow Tape; Weight estimation; Patient safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Accuracy of an algorithm and the Broselow Tape — Computer based comparison of the two devices based on collected patient data

SUMMARY:
The purpose of this prospective single center study is to investigate if a developed algorithm is more accurate than the Broselow Tape (BT). For this study 500 patients are required to collect anonymized data (length, weight, age, anaesthesia material used during anaesthesia) for achieving a power of 80% during statistical analysis. The main hypothesis ist that the algorithm has a better accuracy than the BT.

DETAILED DESCRIPTION:
This prospective single center study is performed at the university children's hospital zurich. Patients planned for surgery in general anaesthesia with intubation, aged 0 to 16 years and with a body length suitable for the emergency tapes can be included in this study. Patient and parental information is performed during the pre-anaesthetic visit.

After written consent the patient will be included. Patient ́s length and weight will be measures earliest one day before data collection. Data collection during anaesthesia has no influence on the daily anaesthesia routine and has no impact on patient safety and anaesthesia. Patient's data is made anonymous for further inspection. Data is documented in Microsoft Excel and statistical analysis calculated with SPSS.

500 patients are needed for a power of 80%. Primary outcome parameter is length- based weight estimation, secondary outcome parameters are length-based age estimation and the correctness of recommended anaesthesia material (endotracheal tube, laryngeal mask, oropharyngeal mask and face mask). Both tools (algorithm and BT) will be compared with each other regarding primary and secondary outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* body length suitable with the investigated emergency tapes
* all patients aged 0 -16 years
* receiving general anaesthesia with intubation or laryngeal mask

Exclusion Criteria:

* Already included in this study once
* missing patient or parental consent

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients planned for elecitve surgery in general anaesthesia
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
length-based weight-estimation by algorithm | during anaesthesia
  The by the algorithm estimated bodyweight based on the patient's Body length is investigated regarding the estimations accuracy and cases in the +/- 10% interval

SECONDARY OUTCOMES:
length based age estimation | during anaesthesia
  The by the algorithm estimated age based on the patient's body length is investigated regarding the estimations accuracy
size of endotracheal tube | during anaesthesia
  The by the algorithm suggested endotracheal tube based on the patient's Body length is investigated regarding the correctness
size of laryngeal mask | during anaesthesia
  The by the algorithm suggested laryngeal mask based on the patient's Body length is investigated regarding the correctness
size of facemask | during anaesthesia
  The by the algorithm suggested facemask based on the patient's body length is investigated regarding the correctness
size of oropharyngeal tube | during anaesthesia
  The by the algorithm suggested oropharyngeal tube based on the patient's Body length is investigated regarding the correctness

CONTACTS AND LOCATIONS:
Locations (1):
- University Childrens Hospital, Zurich, Switzerland